CLINICAL TRIAL: NCT00043758
Title: Multicenter, Randomized, Double-Blind, Placebo Controlled, Efficacy Study on the Effects of Tolvaptan on Left Ventricular Dilatation in Congestive Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-01-232
Record Dates: First submitted 2002-08-13; First posted 2002-08-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
The purpose of this study is to study the effects of tolvaptan on the size and function of the left heart chamber (ventricle) in patients with congestive heart failure (CHF)

ELIGIBILITY:
History of congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2002-07; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Locations (40):
- United States (35):
  - Desert Cardiology of Tucson, Tucson, Arizona
  - Arkansas Heart, Little Rock, Arkansas
  - San Diego Cardiac Center, San Diego, California
  - Northern California Medical Associates, Santa Rosa, California
  - Cardiovascular Consultants Medical Group, Inc., Walnut Creek, California
  - University of Colorado, Denver, Colorado
  - The Hoffman Heart Institute of CT/St. Francis Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Cardiology Associates of Fort Lauderdale, Fort Lauderdale, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Charlotte Heart Group, Port Charlotte, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Cardiovascular Associates of Augusta, PA, Augusta, Georgia
  - Georgia Heart Specialists, Covington, Georgia
  - Illinois Heart and Lung Associates, SC, Normal, Illinois
  - The Care Group, LLC, Indianapolis, Indiana
  - Medical Research Institute, Slidell, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Maine Cardiology Associates, Portland, Maine
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Mystic Cardiology Associates, Inc., Medford, Massachusetts
  - Harper Hospital/Wayne State University, Detroit, Michigan
  - John Dingell VA Medical Center, Detroit, Michigan
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - South Bay Cardiovascular Associates, West Islip, New York
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - North Ohio Research LTD, Lorraine, Ohio
  - North Ohio Research LTD., Sandusky, Ohio
  - Medical College of Pennsylvania, Philadelphia, Pennsylvania
  - Guthrie Clinic, LTD, Sayre, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - University Cardiology Foundation, Providence, Rhode Island
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - Stern Cardiovascular Center, Memphis, Tennessee
- Canada (5):
  - Health Sciences Center, Winnipeg, Manitoba
  - Health Sciences Center Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - London Health Sciences Center, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Toronto Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Udelson JE, McGrew FA, Flores E, Ibrahim H, Katz S, Koshkarian G, O'Brien T, Kronenberg MW, Zimmer C, Orlandi C, Konstam MA. Multicenter, randomized, double-blind, placebo-controlled study on the effect of oral tolvaptan on left ventricular dilation and function in patients with heart failure and systolic dysfunction. J Am Coll Cardiol. 2007 Jun 5;49(22):2151-9. doi: 10.1016/j.jacc.2007.01.091. Epub 2007 May 18. PMID 17543634